CLINICAL TRIAL: NCT05811273
Title: Effects of Physical Readiness Training on Speed, Power, and Dynamic Balance in Badminton Players
Brief Title: Effect of Physical Readiness Training In Badminton Players
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0407
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Sports
Keywords: Badminton player, Physical readiness Training
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physical readiness training (Experimental): Bend and Reach:5 repetitions, Rear Lunge:5 repetitions per leg, High Jumper:5 repetitions, Rower:5 repetitions, Squat Bender:5 repetitions, Windmill:5 repetitions, Forward Lunge:5 repetitions per leg, Prone Row:5 repetitions, Bent-Leg Body Twist:5 repetitions per side, Push-Up:5 repetitions.
  Interventions: Other: physical readiness training
- control group (Active Comparator): general routine exercises
  Interventions: Other: Control group

INTERVENTIONS:
Other: physical readiness training — Bend and Reach:5 repetitions, Rear Lunge:5 repetitions per leg, High Jumper:5 repetitions, Rower:5 repetitions, Squat Bender:5 repetitions, Windmill:5 repetitions, Forward Lunge:5 repetitions per leg, Prone Row:5 repetitions, Bent-Leg Body Twist:5 repetitions per side, Push-Up:5 repetitions.
  Arms: physical readiness training
Other: Control group — general exercises
  Arms: control group

SUMMARY:
Badminton is an extremely demanding sport. At an elite level, players are often required to perform at their limits of speed, agility, flexibility, endurance and strength. On top of all of this, players must maintain a high state of concentration in order to meet the tactical / mental demands of dealing with their opponents. In young badminton players, the most important attributes are high levels of skill. A long-term commitment to endurance training is necessary to reach and maintain a player full physical potential. These are two primary objectives of the endurance program are to prevent injury and enhance the abilities to play the game. Endurance plays the key role in all motor abilities, technical skills and tactical actions. Endurance performance capacity has long been recognized as important prerequisite for on field performance for badminton players.

DETAILED DESCRIPTION:
Badminton is an extremely demanding sport. At an elite level, players are often required to perform at their limits of speed, agility, flexibility, endurance and strength. On top of all of this, players must maintain a high state of concentration in order to meet the tactical / mental demands of dealing with their opponents. In young badminton players, the most important attributes are high levels of skill. A long-term commitment to endurance training is necessary to reach and maintain a player full physical potential. These are two primary objectives of the endurance program are to prevent injury and enhance the abilities to play the game. Endurance plays the key role in all motor abilities, technical skills and tactical actions. Endurance performance capacity has long been recognized as important prerequisite for on field performance for badminton players.

This study will be a randomized controlled trial in which 28 sample size will be taken. The participants will be allocated into control and experimental group. The sample will be taken from Pakistan Sports Board. Control group will follow their daily warm up activities. Interventional group will follow the physical readiness training. Physical readiness training in experimental group adding following exercises along with their conventional exercises. Bend and Reach:5 repetitions, Rear Lunge:5 repetitions per leg, High Jumper:5 repetitions, Rower:5 repetitions, Squat Bender:5 repetitions, Windmill:5 repetitions, Forward Lunge:5 repetitions per leg, Prone Row:5 repetitions, Bent-Leg Body Twist:5 repetitions per side, Push-Up:5 repetitions. And control group population will continue with their conventional exercises only. These exercises will continue for 4 weeks, 3 days per week. Speed (shuttle run test), Power (vertical jump test), Balance (star excretion test). Comparison of two groups control and interventional be done by applying independent sample t-test and p-value < 0.05 will be taken as significance.

ELIGIBILITY:
Inclusion Criteria:

* Males
* 7-30 years of age
* playing experience of at least 1 years and has regular practices

Exclusion Criteria:

* Any recent injury that required medical attention;
* Significant musculoskeletal, neurological, visual, vestibular, cardiorespiratory, or cognitive disorders
* players who worked in occupations involving heavy manual work

Ages: 17 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-03-25 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-22 (Estimated)

PRIMARY OUTCOMES:
Shuttle run test | 4 weeks
  The Interval Shuttle Run Test started directly after the warm-up. Subjects were required to run back and forth on a 20-m course with pylons set 3 m before the turning lines.
Vertical jump test | 4 week
  The Vertical Jump test is used to evaluate a candidate's lower-body strength. A vertical jump test gauge is used to conduct the test. Applicants should stand with their feet level and hip width apart beneath the testing gauge, with their dominant side closer to the gauge. The person then raises their dominant arm and fingers vertically over their head.
  On the test gauge, the test assessor then set the applicant's reach height to zero (0). The leap must be done with both feet flat on the ground without taking a step or running up from the starting position. To safeguard their lower limbs, candidates must take off and land with both feet. Only two (2) tries are permitted for applicants who must leap 30cm or greater
star excursion balance test | 4 week
  The SEBT (Standing Excursion Balance Test) evaluates postural control and dynamic balance. It is currently widely used as a clinical evaluation tool. SEBT necessitates a combination of lower extremity strength, flexibility, and balance. This test is useful in determining whether or not a lower extremity athlete is at danger of injury, as well as musculoskeletal disorders in the lower limb, following a training programmed that improves postural control

CONTACTS AND LOCATIONS:
Overall Officials: Amna Shahid, t-DPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Borad, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No